CLINICAL TRIAL: NCT00819481
Title: Post-Market Study of the 3DKnee™ System Protocol No. PS -- 700
Brief Title: Post-Market Study of the 3DKnee™ System
Status: Completed | Type: Observational
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Sponsor
Other Study IDs: PS - 700
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2017-02

CONDITIONS: Degenerative Joint Disease; Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis
Keywords: Total knee replacement
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 3DKnee: Post Market Study
  Interventions: Device: 3DKnee™ System

INTERVENTIONS:
Device: 3DKnee™ System — Total knee replacement joint for subjects with knee osteoarthritis and willing to participate in the study.

SUMMARY:
The purpose of this study is to evaluate the use and efficacy of the 3DKnee™ System for total knee replacement surgery.

DETAILED DESCRIPTION:
Total knee replacement surgery is widely accepted as effective treatment for degenerative joint disease (DJD), osteoarthritis and rheumatoid arthritis. Relief of patient pain and return of mobility are the primary goals that can be accomplished by this surgery. The purpose of this study is to evaluate the use and efficacy of the 3DKnee™ System for total knee replacement surgery. The study will take place at multiple sites across the United States and be managed by the Encore Medical Clinical Affairs Department. The study will include only patients who meet the indications for use criteria for the 3DKnee™ System and who are candidates for primary knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* This must be a primary knee replacement on this knee.
* Patient is over 18 years of age or older
* Have knee joint disease related to one or more of the following

  * degenerative joint disease, including osteoarthritis or traumatic arthritis
  * Avascular necrosis of the femoral condyles
  * Post-traumatic loss of joint configuration, particularly when there is patellofemoral erosion, dysfunction or prior patellectomy
  * Moderate valgus, varus, or flexion deformities
  * Rheumatoid arthritis
* Patient is likely to be available for evaluation for the duration of the study
* Able and willing to sign the informed consent and follow study procedures
* Patient is not pregnant

Exclusion Criteria:

* Is younger than 18 years of age
* If there has been a total knee replacement on this knee in the past (no revisions allowed in study)
* Infection, or history of infection, acute or chronic, local or systemic
* Alcoholism or other addictions
* Muscular, neurological or vascular deficiencies which compromise the affected extremity
* Obesity
* Insufficient bone quality
* Loss of ligamentous structures
* High levels of physical activity
* Materials sensitivity
* Prisoner
* Mental conditions that may interfere with the patient's ability to give an informed consent or willingness to fulfill the study requirements
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are over 18 years of age and are candidates for a primary total knee replacement.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
efficacy of total knee system | 2 year

SECONDARY OUTCOMES:
change in Knee Society Score | 5 year
change in pain from pre-op to post-op | 5 year
patient satisfaction | 5 year
change in WOMAC Osteoarthritis Index from pre-surgery | 5 year
change in Oxford Knee Score from pre-surgery | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: John W. McAllister, M.D., Principal Investigator — St. Peter's Bone and Joint Surgery; Barry J Waldman, M.D., Principal Investigator — OrthoMaryland
Locations (8):
- United States (8):
  - Longo Orthopedics, Scottsdale, Arizona
  - Center for Excellence, Fresno, California
  - OrthoMaryland, Baltimore, Maryland
  - Metro Orthopedics and Sports Therapy, Silver Spring, Maryland
  - Leslie Orthopedics and Sports Medicine, Camdenton, Missouri
  - St. Peter's Bone & Joint Surgery, City of Saint Peters, Missouri
  - Texas Center for Joint Replacement, Plano, Texas
  - Rimrock Orthopedics, St. George, Utah

REFERENCES:
- See also: Sponsor company home page — http://www.djosurgical.com